CLINICAL TRIAL: NCT06780527
Title: Clinical Performance and Radiographic Assessment of Resin Composite Restoration After Dentin Biomodification by Grape Seed Extract in Vital Teeth With Deep Occlusal Carious Lesions. "18-M Randomized Clinical Trial"
Brief Title: Clinical Performance of Resin Composite Restoration After Dentin Biomodification by Grape Seed Extract in Deep Carious Lesions.
Acronym: GSE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwah Faker Mohammed Al-Emad, Master's student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dentin Biomodification(G.S.E)
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Deep Carious Lesions
Keywords: Deep caries, Partial caries removal, Grape seed extract,
MeSH Terms: interventions — Grape Seed Extract

STUDY DESIGN:
Intervention Model Description: Two parallel arms randomized clinical trial with equal allocation ratio.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Application of resin composite restoration after partial caries removal without application of dentin pretreatment or biomodifier.
- Intervention group (Experimental): Application of resin composite restoration after partial caries removal with application of 15% GSE as dentin pretreatment.
  Interventions: Other: 15% Grape seed extract as dentin pretreatment

INTERVENTIONS:
Other: 15% Grape seed extract as dentin pretreatment — using proanthocyanidin-rich grape seed extract as a biomodifier for dentin improved the mechanical properties of dental collagen by cross-linking and dehydrating fibrils. This made the collagen substrate more suitable for hybridization. It also acted as a non-specific MMP-inhibitor, protecting exposed collagen fibrils from biodegradation from dentin proteases.
  Arms: Intervention group

SUMMARY:
This study will evaluate the clinical and radiographic performance of resin composite restoration after utilized a grape seed extract as dentin biomodification in vital teeth with deep occlusal carious lesions (ICDAS 5-6) after selective soft dentin removal technique.

DETAILED DESCRIPTION:
In dentistry, treating deep carious lesions in vital permanent teeth is one of the most contentious issues. Traditional management of such lesions often compromises the tooth structure and exposes the pulp, necessitating further invasive options such as endodontic treatment. Untreated deep carious lesions can result in significant pain and discomfort. Therefore, certain individuals may decide on tooth extraction rather than undergoing treatment.

The International Caries Consensus Collaboration (ICCC) group strongly recommends selective removal of soft dentine (SRSD) in deep-cavitated lesions that extend into dentin tissue. The one-stage partial caries removal technique involves selective removal to soft dentine (SRSD), which involves removing peripheral carious tissue to firm dentin. This process ensures hermetic sealing of the restoration and leaves a layer of soft carious tissue over the pulp to prevent pulpal exposure.

Recent studies have concentrated on the capacity of medicinal plants and their extracts to remineralize dentin. This process isn't simply a matter of spontaneous precipitation or mineral nucleation but involves the growth of existing crystals within the dentin lesion . Proanthocyanidin-rich grape seed extract (PA-rich GSE) is one promising example that is able to remineralize demineralized dentin, enhance collagen interaction, improve mineral density, preserve collagen matrix, and inhibit matrix metalloproteinases (MMPs) and exhibit low toxicity, making it a suitable candidate for intraoral application.

ELIGIBILITY:
Inclusion Criteria:

* Patient-related criteria:

  1. Adult patients (age: 22-42 years) of both genders.
  2. Good oral hygiene.
  3. Willing to sign the informed consent.
  4. Co-operative patients who accept the follow-up period.
* Tooth-related criteria:

  1. Posterior permanent caries (ICDAS 5&6).
  2. Radiographically, caries is extending 50% of dentine with a radiopaque layer between the carious lesion and the pulp chamber.
  3. Sensible teeth according to cold pulp test.
  4. Negative response in percussion test.

Exclusion Criteria:

* Patient-related criteria:

  1. Allergy to any of the restorative materials.
  2. Patients undergoing orthodontic treatment with fixed appliances.
  3. Pregnant women.
  4. Patients with debilitating systemic diseases.
  5. Patient who frequently use analgesic or any drugs that could mask the pain.
* Tooth-related criteria:

  1. Teeth with previous restorations.
  2. Spontaneous pain or prolonged pain (more than 15 s) after sensitivity test (cold test), which would indicate irreversible pulpitis.
  3. Negative sensibility tests, periapical radiolucencies and sensitivity to axial or lateral percussion.
  4. Mobile teeth, indicating periodontal disease or trauma.
  5. External or internal resorption.
  6. Chipped teeth or Cuspal loss

Ages: 22 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Performance (Biological properties), Revised FDI criteria. (Clinically excellent-Success rate) | 18 month
  Postoperative hypersensitivity and pulpal status/ Caries at restoration margins (CAR), Scores
  1. clinically very good
  2. clinically good
  3. clinically sufficient
  4. clinically unsatisfactory
  5. clinically poor

SECONDARY OUTCOMES:
Radiographic Assessment, Digital radiography | 18 month
  Greyscale values ranged from 0 (black pixel) to 255 (white pixel).

CONTACTS AND LOCATIONS:
Overall Officials: Pro. Heba Salah El Din Hamza (H.H.) Head of Conservative Dentistry Department, Cairo University., Professor, Study Director — Professor, Conservative Dentistry Department, Faculty of Dentistry, Cairo University, Egypt.; Dr. Rawda Hesham Abd ElAziz (R.H.) Lecturer of Conservative Dentistry Department,Cairo University, Lecturer, Study Director — Lecturer of Conservative Dentistry Department, Faculty of Dentistry, Cairo University, Egypt.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Kls N, Ramar K. Evaluation of the Genotoxic Effects of Grape Seed Extract and Marine Collagen Peptide on the Fibroblast Cell Line: An In Vitro Study. Cureus. 2024 Jun 3;16(6):e61605. doi: 10.7759/cureus.61605. eCollection 2024 Jun. PMID 38962594
- [Result] Hickel R, Mesinger S, Opdam N, Loomans B, Frankenberger R, Cadenaro M, Burgess J, Peschke A, Heintze SD, Kuhnisch J. Revised FDI criteria for evaluating direct and indirect dental restorations-recommendations for its clinical use, interpretation, and reporting. Clin Oral Investig. 2023 Jun;27(6):2573-2592. doi: 10.1007/s00784-022-04814-1. Epub 2022 Dec 12. PMID 36504246
- [Result] Gozetici-Cil B, Erdem-Hepsenoglu Y, Tekin A, Ozcan M. Selective removal to soft dentine or selective removal to firm dentine for deep caries lesions in permanent posterior teeth: a randomized controlled clinical trial up to 2 years. Clin Oral Investig. 2023 May;27(5):2125-2137. doi: 10.1007/s00784-022-04815-0. Epub 2022 Dec 3. PMID 36460919
- [Result] Cushley S, Duncan HF, Lundy FT, Nagendrababu V, Clarke M, El Karim I. Outcomes reporting in systematic reviews on vital pulp treatment: A scoping review for the development of a core outcome set. Int Endod J. 2022 Sep;55(9):891-909. doi: 10.1111/iej.13785. Epub 2022 Jun 30. PMID 35704241
- [Result] Bedran-Russo AK, Castellan CS, Shinohara MS, Hassan L, Antunes A. Characterization of biomodified dentin matrices for potential preventive and reparative therapies. Acta Biomater. 2011 Apr;7(4):1735-41. doi: 10.1016/j.actbio.2010.12.013. Epub 2010 Dec 16. PMID 21167964
- [Result] Balalaie A, Rezvani MB, Mohammadi Basir M. Dual function of proanthocyanidins as both MMP inhibitor and crosslinker in dentin biomodification: A literature review. Dent Mater J. 2018 Mar 30;37(2):173-182. doi: 10.4012/dmj.2017-062. Epub 2017 Nov 23. PMID 29176304
- [Result] Anumula L, Ramesh S, Kolaparthi VSK, Kirubakaran R, Karobari MI, Arora S, Saleh AA, Aldowah O, Messina P, Scardina GA. Role of Natural Cross Linkers in Resin-Dentin Bond Durability: A Systematic Review and Meta-Analysis. Materials (Basel). 2022 Aug 17;15(16):5650. doi: 10.3390/ma15165650. PMID 36013786
- [Result] Abd ElAziz RH, Ragab RA, Elzayat GA. Comparative evaluation and patient satisfaction with an electrical impedance-based device versus digital radiography in the estimation of remaining dentin thickness in carious posterior permanent teeth: (Diagnostic accuracy study). BMC Oral Health. 2024 Apr 8;24(1):429. doi: 10.1186/s12903-024-04205-w. PMID 38584280